CLINICAL TRIAL: NCT01857271
Title: EValuation of Erlotinib as a Neoadjuvant Therapy in Stage III NSCLC Patients With EGFR Mutations (EVENT Trial)
Brief Title: Erlotinib Hydrochloride Before Surgery in Treating Patients With Stage III Non-Small Cell Lung Cancer
Acronym: EVENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Haiying Cheng, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-233; NCI-2013-02219 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-233-004; 2013-233 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (erlotinib hydrochloride and thoracotomy) (Experimental): Patients receive erlotinib hydrochloride PO QD for 2 months and then undergo thoracotomy.
  Interventions: Drug: Erlotinib Hydrochloride; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774
Procedure: Therapeutic Conventional Surgery — Undergo thoracotomy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well erlotinib hydrochloride works before surgery in treating patients with stage III non-small cell lung cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erlotinib hydrochloride before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of mediastinal nodal clearance and complete pathological response after neoadjuvant erlotinib (erlotinib hydrochloride) in patients with epidermal growth factor receptor (EGFR) mutated stage III non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To determine the progression free survival in patient population of EGFR mutated stage III NSCLC patients who are treated with neoadjuvant erlotinib therapy.

II. To determine the overall survival. III. To estimate the overall response rate from neoadjuvant erlotinib. IV. To estimate the surgical resection rate. V. To evaluate the safety of neoadjuvant erlotinib.

TERTIARY OBJECTIVES:

I. To determine several molecular and cellular biomarkers in the tumors, the skin and the serum that are predictive of the efficacy of neoadjuvant erlotinib.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) for 2 months and then undergo thoracotomy.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven (either histologic or cytologic) diagnosis of stage IIIA or IIIB non-small cell lung cancer; (according to American Joint Committee on Cancer [AJCC] staging, 7th edition) within 4 weeks of registration; the patient should have histologically or cytologically confirmed N2 disease
* Activating mutation in EGFR
* No prior chemotherapy or radiation for lung cancer
* Patients may be potentially resectable or unresectable
* Stage III A or B disease, including no distant metastases- based on following diagnostic workup:

  * History/physical examination prior to registration
  * Computed tomography (CT) scan of the chest or positron emission tomography (PET) scan within 28 days of study entry
  * CT scan of abdomen or magnetic resonance imaging (MRI) of abdomen or PET scan within 28 days of study entry
  * An MRI of the brain or head CT scan with contrast within 28 days of study entry
  * Total body PET scan within 28 days of study entry
  * Mediastinoscopies are highly recommended
* Patients must have measurable or evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500 cells/ul
* Platelets >= 100,000 cells/ul
* Hemoglobin >= 9.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= g/dl is acceptable)
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin < 2.0 times the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x the ULN
* Women of childbearing potential must have:

  * A negative serum or urine pregnancy test (sensitivity =< 25 IU human chorionic gonadotropin [HCG]/L) within 72 hours prior to the start of study drug administration
  * Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy
* Ability to take oral medication
* Patient must sign study specific informed consent prior to study entry

Exclusion Criteria:

* Pleural or pericardial effusion

  * Pleural effusions allowed if one of the following conditions are met: 1) negative cytology after adequate sampling by thoracentesis 2) effusion seen on CT scan but not on chest x-ray and deemed too small to tap under CT or ultrasound guidance
* Severe, active co-morbidity, defined as follows:

  * Cardiac symptoms; any of the following should be considered for exclusion:

    * Uncontrolled angina, congestive heart failure or myocardial infarction (MI) within (6 months)
    * Diagnosed congenital long QT syndrome
    * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
    * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec)
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (=< 3 months) significant gastrointestinal bleeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
* Men and women who:

  * Are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or women who:

    * Have a positive pregnancy test at baseline, or
    * Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haiying Cheng, Principal Investigator — Albert Einstein College of Medicine
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were enrolled on 11/7/2013, 5/2014, and 9/24/2014.
Pre-assignment Details: The study was difficult to enroll and eventually terminated/closed.
Groups:
- Treatment (Erlotinib Hydrochloride): Patients receive erlotinib hydrochloride PO QD for 2 months and then undergo restaging procedures to evaluate for surgery.
  Erlotinib Hydrochloride: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Erlotinib Hydrochloride)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Erlotinib Hydrochloride and Thoracotomy)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Two females, one male.
  Participants
    Female | 2
    Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Mediastinal Nodal Clearance, Defined as Pathologically Negative N2 Disease in the Final Surgical Resection Specimen or Mediastinoscopy
Time Frame: 3 years 9 months
Population: The study was closely prematurely due to poor accrual. No final analysis was performed due to very low number of subjects.
Arm/Group | Treatment (Erlotinib Hydrochloride and Thoracotomy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment (Erlotinib Hydrochloride and Thoracotomy)
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erlotinib Hydrochloride and Thoracotomy) (N=3)
Diarrhea (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT01857271/Prot_SAP_000.pdf